CLINICAL TRIAL: NCT03841409
Title: Peak Plasma Levels of Bupivacaine After an Erector Spinae Block
Brief Title: Peak Plasma Levels of Bupivacaine After an Erector Spinae Block (ESP)
Status: Completed | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Other Study IDs: 18.308
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2021-07

CONDITIONS: Pharmacokinetics; Anesthesia, Local

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bupivacaine dosage in ESP block: The pharmacokinetics of bupivacaine 0.5% with epinephrine 5 mcg/mL for a total dose of 2mg/kg of ideal body weight following an ESP block will be determined by the collection of blood samples at predetermined time points.
  Interventions: Other: Collection of blood samples

INTERVENTIONS:
Other: Collection of blood samples — Nine blood samples will be collected to determine bupivacaine pharmacokinetics at T10min, T20min, T30min, T45min, T60min, T90min, T120min, T180min, and T240min. T0 will be defined as the end of bupivacaine injection.

SUMMARY:
The primary objective of the study is to measure plasma levels of bupivacaine following erector spinae (ESP) regional block in patients undergoing mastectomy.

DETAILED DESCRIPTION:
Breast cancer is one of the most frequent types of cancer in women. Mastectomy is important in treating these cases; however, sometimes it is associated with acute and chronic pain. Multimodal analgesia, combining drug therapy and regional anesthesia, can help in preventing acute and perhaps chronic pain in breast cancer patients undergoing mastectomy.

Erector spinae block is a new regional anesthesia technique that has emerged to treat thoracic pain following thoracic and breast surgery. It consists of injecting local anesthetics in the space located between the erector and paravertebral muscles using ultrasound guidance. The injection can be done at the level of T5 allowing distribution of the drug to upper and lower dermatomes.

The dose of local anesthetic injected after erector spinae block should aim to maximize analgesia while minimizing the chance of toxic systemic concentrations. Defining the rate of absorption of local anesthetics into the blood after an erector spinae block will therefore help anesthesiologists determinate optimal analgesic doses, in terms of both safety and effectiveness.

This observational study will determine bupivacaine pharmacokinetics after single shot erector spinae block with bupivacaine, to further define the right dose and duration of surveillance in post-anesthesia care.

Methods:

For the erector spinae block, the patient will be placed in the sitting position. Using an ultrasound machine with a high frequency linear probe (Sonosite, HFL50 15-6MHz) placed in the parasagittal plane, 3cm away from the midline, the anesthesiologist will position an insulated hyperechoic needle (50-80 mm, 22 gauge, SonoPlex STIM, Nanoline, Pajun, Germany) at the level of the 5th thoracic vertebrae, between the erector spinae and the paravertebral muscles. The anesthesiologist will confirm the correct position of the needle with the injection of 1 mL of 5% dextrose. Then, after negative aspiration, he will inject bupivacaine 0.5% with epinephrine 5 mcg/mL in 5 ml aliquots for a total dose of 2mg/kg of ideal body weight (maximum of 150mg).

The end of injection will be considered as T0. Collection of 4.5mL of blood will be performed at T10min, T20min, T30min, T45min, T60min, T90min, T120min, T180min, and T240min.

Blood tubes will be immediately placed on ice to be ultimately sent to the laboratory for centrifugation and measurement of bupivacaine level using liquid chromatography-tandem mass spectrometry (LC-MS/MS) for each of the samples.

General anesthesia will then be induced in the operating room with no additional bupivacaine allowed by the anesthesiologist or the surgeon. After surgery, in the Post-Anesthesia Care Unit, the level of the sensory block will be identified by pinprick and the quality of analgesia will be evaluated using a verbal numerical rating scale, and opioid consumption will be noted.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Undergoing unilateral mastectomy under erector spinae block and general anesthesia

Exclusion Criteria:

* Patient's refusal or inability to consent
* Allergy, hypersensibility or resistance to local anesthetic
* Contra-indication to regional anesthesia: infection in the designated area, acquired or congenital coagulopathy
* Severe hepatic or renal insufficiency (GFR<30 mL/min)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing unilateral mastectomy under general anesthesia and erector spinae block for post-operative pain management.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2019-10-16 (Actual)

PRIMARY OUTCOMES:
Maximal plasma concentration (Cmax) of bupivacaine after erector spinae block | The end of injection of bupivacaine will be considered as T0. Blood samples at T10, T20, T30, T45, T60, T90, T120, T180, and T240minutes will be collected to further analyze plasmatic bupivacaine values at these timepoints.
  The Cmax will be estimated by interpolation based on the plasmatic bupivacaine values obtained after the analysis of the blood samples.

SECONDARY OUTCOMES:
Time (Tmax) to maximum plasma concentration Cmax of bupivacaine | The end of injection of bupivacaine will be considered as T0. Blood samples at T10, T20, T30, T45, T60, T90, T120, T180, and T240minutes will be performed to further analyze plasmatic bupivacaine values at these timepoints.
  The Tmax will be estimated by interpolation based on the plasmatic bupivacaine values obtained after the analysis of the blood samples.
Sensory block level 30 minutes after arriving to Post-Anesthesia Care Unit | 30 minutes after arriving to Post-Anesthesia Care Unit
  Sensory block level will be measured with a 6.1g von Frey filaments.
Post-operative pain using verbal numerical rating scale | 30 minutes after arriving to Post-Anesthesia Care Unit
  The quality of postoperative analgesia at rest will be evaluated with a verbal numeric scale (VNS) where 0 represents 'no pain' and 10 represents 'the worst pain'.
Total opioid dose needed during Post-Anesthesia Care Unit stay (PACU) | After the surgery, from the entry in the Post-Anesthesia Care Unit to the discharge from the Post-Anesthesia Care Unit, for an average of one-hour stay.
  The total dose of opioids used by the patients during the PACU stay will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Williams, MD, PhD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided